CLINICAL TRIAL: NCT06688435
Title: A Phase I Study to Evaluate BCMA-targeted Chimeric Antigen Receptor T Cell (SYS6020 Injection) in Patients With Refractory Generalized Myasthenia Gravis
Brief Title: A Study to Evaluate the Safety and Preliminary Efficacy of SYS6020 CAR T-cells in Patients With Refractory Generalized Myasthenia Gravis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SYS6020-004
Record Dates: First submitted 2024-11-06; First posted 2024-11-14 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Intervention Model Description: This is an open-label, two-phase (dose-escalation and dose-expansion), multicenter, phase I clinical study. The dose-escalation phase adopts a sequential design model, including 5 arms for 5 dose level. The arms of dose-expansion phase depends on the number of recommended dose, which may be 1-2 recommended dose.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- SYS6020 injection: 2*106CAR+ T-cells per kg(dose level 1) (Experimental): Participants will undergo leukapheresis to isolate peripheral blood mononuclear cells to manufacture SYS6020 injection, during which no lymphodepleting chemotherapy will be performed. Participants will receive 3 doses treatment of SYS6020 injection, with a dose level of 2*106CAR+ T-cells per kg. If one DLT occurs in three participants, additional 3 ones may be considered to be enrolled after SMC safety data review and make a determination.
  Interventions: Biological: SYS6020 injection
- SYS6020 injection: 6*106CAR+ T-cells per kg(dose level 2) (Experimental): Participants will undergo leukapheresis to isolate peripheral blood mononuclear cells to manufacture SYS6020 injection, during which no lymphodepleting chemotherapy will be performed. Participants will receive 3 doses treatment of SYS6020 injection, with a dose level of 6*106CAR+ T-cells per kg. If one DLT occurs in three participants, additional 3 ones may be considered to be enrolled after SMC safety data review and make a determination.
  Interventions: Biological: SYS6020 injection
- SYS6020 injection: 1.8*107CAR+ T-cells per kg(dose level 3) (Experimental): Participants will undergo leukapheresis to isolate peripheral blood mononuclear cells to manufacture SYS6020 injection, during which no lymphodepleting chemotherapy will be performed. Participants receive 3 doses of SYS6020 injection, with a dose level of 1.8*107CAR+ T-cells per kg. If one DLT occurs in three participants, additional 3 ones may be considered to be enrolled after SMC safety data review and make a determination.
  Interventions: Biological: SYS6020 injection
- SYS6020 injection: 3.6*107CAR+ T-cells per kg(dose level 4) (Experimental): Participants will undergo leukapheresis to isolate peripheral blood mononuclear cells to manufacture SYS6020 injection, during which no lymphodepleting chemotherapy will be performed. Participants receive 3 doses of SYS6020 injection, with a dose level of 3.6*107CAR+ T-cells per kg. If one DLT occurs in three participants, additional 3 ones may be considered to be enrolled after SMC safety data review and make a determination.
  Interventions: Biological: SYS6020 injection
- SYS6020 injection: 5.4*107CAR+ T-cells per kg(dose level 5) (Experimental): Participants will undergo leukapheresis to isolate peripheral blood mononuclear cells to manufacture SYS6020 injection, during which no lymphodepleting chemotherapy will be performed. Participants receive 3 doses of SYS6020 injection, with a dose level of 5.4*107CAR+ T-cells per kg. If one DLT occurs in three participants, additional 3 ones may be considered to be enrolled after SMC safety data review and make a determination.
  Interventions: Biological: SYS6020 injection

INTERVENTIONS:
Biological: SYS6020 injection — The SYS6020 is an injection of autologous CAR-T cells that have been temporarily transfected with LNP-mRNA targeting BCMA. Before each dosing, the infusion eligibility of SYS6020 is assessed by the investigator, and the eligible participants will receive 3 dosing SYS6020 injection treatment. The dosing interval is 7 days according to the protocol design.

SUMMARY:
This study is a single-arm, open, 2-stage (dose-escalation phase and dose-expansion phase), multi-center, phase I clinical trial to evaluate the safety and tolerance of SYS6020 injection in the participants with refractory systemic myasthenia gravis, and determine the recommended dose (RD) for subsequent studies of the product, and to preliminarily evaluate the clinical efficacy of the product, as well as to explore the pharmacokinetics and immunogenicity of the product in vivo.

The dose-escalation phase and dose-expansion phase include 7 periods, and they are respectively in sequence as follows: the screening period, apheresis period, pre-dosing assessment, SYS6020 injection infusion, DLT observation period, the primary follow-up period (6 months), and the long-term follow-up period (5 years). The DLT observation period is 28 days after receiving SYS6020 injection. The participants will not undergo lymphodepleting chemotherapy.

The efficacy and safety profile of the participants will be continuously assessed during the trial. Efficacy measurement includes the MG-ADL, QMG, MGC, MG-QoL 15R scale, MGFA clinical classification, and MGFA post-intervention state (MGFA PIS) grading scales, as well as self-antibodies, etc. Safety measurement includes vital signs, physical examination, laboratory tests, cytokines, and ECG, etc. The adverse events and concomitant therapy will be continuously collected during the trial. In addition, during the study period, blood samples will be collected from participants who have received SYS6020 treatment for PK/PD test, and immunogenicity test.

For the dose-escalation phase, 3 to 5 dose levels are proposed to be explored. The Safety Monitoring Committee (SMC) will discuss the safety data and make a decision if the next SYS6020 injection could be initiated or dose-escalation could be initiated. After the completion of the dose-escalation phase, the recommended doses would be determined for dose-expansion phase. For the dose-expansion phase, further safety and efficacy data will be collected among the participants who will receive the recommended dose of SYS6020 injection.

ELIGIBILITY:
Inclusion Criteria:

* 1) The ages ≥18 and ≤ 65 years old;
* 2)Diagnosed as generalized myasthenia gravis (GMG), the clinical classification of MGFA II-IV；
* 3) Diagnosed as refractory myasthenia gravis (refractory MG) ；
* 4) QMG score >11 in the screening period and before apheresis;
* 5) Positive acetylcholine receptor antibody (AChR-Ab) and/or muscle-specific receptor tyrosine kinase (MuSK) antibody in the screening period;
* 6) The daily dose of concomitant glucocorticoid therapy must not exceed 40mg prednisone or equivalent dose and the dose have to be stable for ≥4 weeks prior to baseline.
* 7) Participants have a thorough understanding of this clinical trial and voluntarily sign a written informed consent form.

Exclusion Criteria:

* 1) Have been known to have allergic reactions, hypersensitivity, intolerance or contraindications to SYS6020（including its active ingredient and excipient dextran 40） or the drugs potentially used in the study, or who have had a previous history of severe allergic reactions;
* 2) Participants with major chronic diseases that are not well-controlled and considered to increase the participant's risk potentially by the investigator;
* 3) Participants with other autoimmune diseases that require systemic treatment. Participants with stable autoimmune thyroid diseases who have a normal thyroid function and are at a stable therapeutic dose are allowed to be enrolled.
* 4) Participants with a severe recurrent infection during the screening period, or any active infection that the investigator considers may affect the patient's participation;
* 5)Participants with a history of positive HIV; participants with positive HBsAg; participants with positive HBcAb and with HBV-DNA above the measurable limit;
* 6) Participants with a history of malignant tumors within the past 5 years or with current active malignant tumors. Participants with successfully treated localized tumors, as well as those with thymomas classified as A, AB and B1 subtypes according to the WHO pathological classifications, are allowed to be enrolled;
* 7) Any serious respiratory system disease.
* 8) Participants with a history of serious cardiovascular disease, such as severe cardiac rhythm or conduction abnormalities.
* 9) Abnormal laboratory findings with clinical significance, including ALT, AST>3*ULN； Scr>1.5*ULN； INR>1.5*ULN, and so on. .
* 10) Individuals with potential disease conditions (including laboratory abnormalities) which are considered of clinical significance by the investigator; individuals with alcohol dependence or drug abuse .
* 11) Individuals with a current psychotic disorder that interferes with adherence.
* 12) Participants with a history of primary immunodeficiency disease, organ or hematopoietic stem cell/bone marrow transplantations before screening; or those planning to undergo a transplantation during the trial;
* 13) Participants with a history of ≥ Grade 2 (CTCAE 5.0 standard) bleeding within 30 days before screening, or those requiring long-term continuous treatments with anticoagulant drugs.
* 14) Participants who have received any CAR-T therapy or gene therapy before.
* 15) Participants who have received intravenous injection of human immunoglobulin (IVIG) or plasmapheresis (PE), plasma separation, or hemodialysis within 1 month before apheresis.
* 16) Participants who have used calcineurin inhibitors, or cyclophosphamide or neonatal Fc receptor antagonists within 3 weeks before apheresis and 8 weeks before the first dosing. Participants who have used targeted B-cell biological agents such as rituximab within 3 months before apheresis. Participants who started receiving eculizumab treatment within 8 weeks before the first dosing；
* 17) Any situations that the investigator believes that the participant is not suitable for this clinical trial for any other reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2033-05-01 (Estimated)

PRIMARY OUTCOMES:
The frequency and the grade of DLT and the incidence of adverse events and serious adverse events. (For the dose-escalation phase) | 12 months
  For the dose-escalation phase, the primary objective is to evaluate the safety of SYS6020, as measured by the frequency and nature of Dose-limiting toxicity (DLT) and the incidence of all adverse events and serious adverse events. DLT is defined as any adverse event related to SYS6020 that occurs within 28 days after the infusion of SYS6020 and that meets certain criteria.
Response rate at 12 months after dosing （For the dose-expansion phase) | 12months
  Response rate is defined as:
  1. The score of Myasthenia Gravis Activities of Daily Living Scale (MG-ADL) and Quantitative Myasthenia Gravis score (QMG) is decreased by ≥2 points from baseline to 12 months after dosing; or
  2. The score of Myasthenia Gravis Composite Scale (MGC) is decreased by ≥3 points from baseline to 12 months after dosing; or
  3. The concentration of specific autoantibodies (i.e., AChR-Ab or MuSK-Ab) is decreased by ≥50% from baseline to 12 months after dosing.

SECONDARY OUTCOMES:
The proportion of MG-ADL score sdecline≥2 | 6 months, 12 months
  The proportion of participants achieving a decline of 2 points or more in MG-ADL from baseline to 6 months and 12 months after dosing (as dose-escalation phase endpoints only); The proportion of participants achieving a decline of 2 points or more in MG-ADL from baseline to 6 months after dosing (as dose-expansion phase endpoints only)
the proportion of QMG score decline≥2 | 6 months, 12 months
  The proportion of participants achieving a decline of 2 points or more in QMG from baseline to 6 months and 12 months after dosing (as dose-escalation phase endpoints only); The proportion of participants achieving a decline of 2 points or more in QMG from baseline to 6 months after dosing (as dose-expansion phase endpoints only)
The proportion of MGC score decline≥3 | 6 months, 12 months
  The proportion of participants achieving a decline of 3 points or more in MGC from baseline to 6 months and 12 months after dosing (as dose-escalation phase endpoints only); The proportion of participants achieving a decline of 3 points or more in MGC from baseline to 6 months after dosing (as dose-expansion phase endpoints only)
The mean change of MG-ADL score | 6 months, 12 months
  the mean change of MG-ADL score from baseline to 6 months and 12 months after dosing (as two-phase joint-endpoints)
The mean change of QMG score | 6 months, 12 months
  the mean change of QMG score from baseline to 6 months and 12 months after dosing (as two-phase joint-endpoints)
The mean change of MG QoL-15R score | 6 months, 12 months
  the mean change of MG QoL-15R from baseline to 6 months and 12 months after dosing (as two-phase joint-endpoints)
The mean change of MGC score | 6 months, 12 months
  the mean change of MGC from baseline to 6 months and 12 months after dosing (as two-phase joint-endpoints)
The mean change of MGFA clinical classification | 6 months, 12 months
  the mean change of MGFA clinical classification from baseline to 6 months and 12 months after dosing (as two-phase joint-endpoints)
The mean change of MGFA PIS grading | 6 months, 12 months
  the mean change of MGFA PIS grading from baseline to 6 months and 12 months after dosing (as two-phase joint-endpoints)
The mean change of hand grip strength | 6 months, 12 months
  the mean change of hand grip strength from baseline to 6 months and 12 months after dosing (as two-phase joint-endpoints)
The mean change of vital capacity | 6 months, 12 months
  the mean change of vital capacity from baseline to 6 months and 12 months after dosing (as two-phase joint-endpoints)
The proportion of participants with concentration titer change of myasthenia gravis-specific autoantibody | 12 weeks
  the proportion of participants whose AChR-Ab or MuSK-Ab concentrations titer is declined by ≥50% from baseline to 12 weeks after dosing (as two phase joint-endpoints)
The incidence of AE and SAE | 12 months
  the incidence of all the adverse events (AE) and serious adverse events (SAE) during 12 months after dosing. (as two phase joint-endpoints)
the pharmacokinetic parameters of SYS6020 injection | 12 months
  the concentrations and pharmacokinetic parameters of SYS6020 CAR+ cells, as well as the gene copies of CAR targeting BCMA.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital, Shandong University, Jinan, China

IPD SHARING:
Plan to Share IPD: No